CLINICAL TRIAL: NCT00440973
Title: Phase II Study of Interleukin- 2 and Bevacizumab in Patients With Progressive Metastatic Renal Cell Carcinoma
Brief Title: Safety Study of Specific Tumor Target Drug Plus Immune System Therapy in Patients With Kidney Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: contract issues
Sponsor: The Methodist Hospital Research Institute (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PAC IRB #03-0194-05; 16117 (Other: Principal Investigator)
Record Dates: First submitted 2007-02-23; First posted 2007-02-27 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Carcinoma, Renal Cell
Keywords: kidney cancer; M3thodist
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — Bevacizumab; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- treatment arm (Other): PI relocated, currently data is no longer available
  Interventions: Drug: Bevacizumab; Drug: Interleukin-2

INTERVENTIONS:
Drug: Bevacizumab — monoclonal antibody with anti-angiogenesis properties used as chemotherapy
  Other Names: Avastin
Drug: Interleukin-2 — immunotherapy - cytokine signaling molecule used as an immune system regulator to trigger T & B lymphocyte proliferation
  Other Names: IL-2

SUMMARY:
The purpose of this study is to determine if the combination of therapy to strengthen the immune system (Interleukin - 2) plus a specific tumor target therapy (Bevacizumab) can prolong the time between the start of treatment and disease progression, decrease tumor size, as well as determine if the combination therapy is safer and less toxic than the standard treatment for renal cell carcinoma.

DETAILED DESCRIPTION:
The standard first-line treatment for patients with metastatic RCC is IL-2 at higher doses, but associated with higher frequency of toxicities. IL-2 given at lower doses have demonstrated similar results than higher doses but it requires further study. RCC is highly vascular and expresses high levels of VEGF. Bevacizumab is a monoclonal antibody directed against the Vascular Endothelial Growth Factor (VEGF) responsible for angiogenesis.

The study is designed to evaluate a response defined as time to progression, safety and toxicity in patients with metastatic renal cell carcinoma. Tissue correlation to evaluate the impact of vascular VEGF on clinical outcome will be retrospectively performed

ELIGIBILITY:
Inclusion Criteria:

* Pathological proof of clear cell carcinoma (or mixed tumors ≥ 75% clear cell component)
* Evidence of measurable metastatic disease, no progression diseases or the patient's condition will not need radiotherapy in the next 4 weeks.
* Previous definitive radiotherapy to 1 metastatic site is acceptable
* At least 4 weeks have elapsed since radiation therapy
* Patients must be free of serious co-morbidity and have a life expectancy of ≥24 weeks
* Patients should have adequate physiologic reserves as evidence of adequate performance status, blood parameters, hepatic and kidney function, no evidence of active cardiac diseases and showing an acceptable function and adequate coagulation profile.

Exclusion Criteria:

* History of central nervous System metastases
* Known HIV positive
* Recent history of brain's vascular disease within 6 months; patients requiring regular antianginal therapy (coronary disease) or insufficient circulation in lower extremities are not eligible
* Active autoimmune disease
* Patients who have had steroid therapy in the past three weeks
* Patients taking concurrent anticancer drugs
* Biphosphonates (Zometa) are not allowed, unless started 4 weeks prior to participation in the study
* Female patients pregnant or breast-feeding
* The patient has an unstable medical condition, such as uncontrolled Diabetes mellitus or Hypertension; active infections requiring systemic antibiotics, antivirals, or antifungal; clinical evidence of cardiac or pulmonary dysfunction including, uncontrolled arrhythmias, unstable coagulation disorders; or recent myocardial infarction (within 6 months)
* Any condition including abnormal laboratory results, that in the opinion of the investigator places the patient at an unacceptable risk if he/she participate in the study
* Prior malignancy (within the last 3 years), except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer or other cancer for which the patient has been - free for at least 3 years
* Uncontrolled Blood pressure > 150/100
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0, anticipation of need for major surgical procedure during the course of the study
* Minor surgery 7 days before day 0
* Serious, non healing wound, ulcer, or bone fracture; and,inability to accomplish the treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2006-10; Primary Completion 2007-10 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
time to progression | During study (currently data no longer available)
  currently data no longer available

SECONDARY OUTCOMES:
Collect data on tumor responses produced by interleukin-2 and Bevacizumab | During study (currently data no longer available)
  currently data no longer available
Evaluate safety and toxicity of the combination of interleukin-2 and Bevacizumab for patients with progressive metastatic renal cell carcinoma. | During study (currently data no longer available)
  currently data no longer available

CONTACTS AND LOCATIONS:
Overall Officials: Robert J. Amato, D.O., Principal Investigator — Baylor College of Medicine - Methodist Hospital
Locations (1):
- Baylor College of Medicine - Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No